CLINICAL TRIAL: NCT06557421
Title: De-Escalation Study Evaluating Venetoclax and Azacitidine Discontinuation in AML Responding Patients
Acronym: STOP VEN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STOP VEN-IPC 2024-001
Record Dates: First submitted 2024-08-09; First posted 2024-08-16 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VEN-AZA de-escalation (Experimental): VEN-AZA de-escalation
  Interventions: Drug: Venetoclax; Drug: Azacitidine

INTERVENTIONS:
Drug: Venetoclax — complete discontinuation of Venetoclax
Drug: Azacitidine — complete discontinuation of Azacitidine

SUMMARY:
The goal of this clinical trial is to test efficacy and safety of a VENETOCLAX-AZACITIDINE (VEN-AZA) de-escalation strategy in Acute Myeloid Leukemia responding patients. The main objectives of the study are:

* Evaluation of the efficacy of VEN-AZA de-escalation strategy by measuring the effect of VEN-AZA discontinuation in term of Disease-Free Survival.
* Evaluation of the other efficacy parameters and safety of VEN-AZA de-escalation strategy.

Patients from the prospective study will be compared to a retrospective cohort of patients who will be selected on the basis of identical eligibility criteria.

Participants will:

* Stop VEN-DASA treatment
* Be closely monitored by regular evaluation of the disease

ELIGIBILITY:
Inclusion Criteria:

1. Female/Male ≥ 18 years of age;
2. Diagnosis of previously untreated AML according to the 2022 International Consensus Classification of Myeloid Neoplasms and Acute Leukemias;
3. VEN-AZA given as first-line treatment;
4. Duration of VEN-AZA therapy of 12 months (+/- 28 days), regardless of duration of VEN-AZA cycles and the doses;
5. Patients in first composite complete remission (CRc) defined as complete remission (CR) or CR with incomplete hematologic recovery (CRi) or CR with partial hematologic recovery (CRh);
6. Absence of detectable minimal residual disease (MRD) performed locally (i.e. MRDneg defined as MCF MRD <0.1% of CD45 expressing cells with the target immunophenotype in bone marrow, or NPM1 or RUNX1-RUNX1T1 or CBFB-MYH11 MRD copy numbers <0.1% in the blood);
7. ECOG <3;
8. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule;
9. Affiliated to the French Social Security or beneficiary of such a health Insurance;
10. Signed informed consent.

Non inclusion Criteria:

1. VEN-AZA given as salvage therapy;
2. Prior allogeneic stem cell transplant;
3. Discontinuation of treatment because of absence or loss of response;
4. Patient in emergency situation or unable to give consent;
5. Severe medical or mental condition precluding the follow up procedures after treatment discontinuation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-12 (Estimated); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival, measured from inclusion (VEN-AZA de-escalation) to the date of morphologic or measurable residual disease relapse or death from any cause, whichever occurs first. | 24 months

SECONDARY OUTCOMES:
Absolute duration of hematologic response, defined as the time from inclusion to relapse or death. | 24 months
Absolute duration of negative measurable residual disease response, defined as the time from inclusion to measurable residual disease relapse or death. | 24 months
Cumulative incidence of relapse, defined as the probability of relapse over time. | 24 months
Overall survival, defined as the time from inclusion (VEN-AZA de-escalation) to death. | 24 months
Second complete remission occurence. | 24 months
Time to second remission, defined as the time between date of treatment re initiation and complete remission. | 24 months
Hospitalization rate associated with VEN-AZA de-escalation. | 24 months
Transfusion occurrence associated with VEN-AZA de-escalation. | 24 months
Grade 3-4 adverse events occurence associated with VEN-AZA de-escalation. | 24 months
Correlation between age and duration of response and survival after VEN-AZA de-escalation. | 24 months
Correlation between FAB classification and duration of response and survival after VEN-AZA de-escalation. | 24 months
Correlation between cytogenetic and molecular alterations and duration of response and survival after VEN-AZA de-escalation. | 24 months
Correlation between number of prior VEN-AZA cycles and duration of response and survival after VEN-AZA de-escalation. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain GARCIAZ, MD PhD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli-Calmettes, Marseille, France

IPD SHARING:
Plan to Share IPD: No